CLINICAL TRIAL: NCT07119502
Title: Implementation of a Minimal Equipment Exercise Intervention in Community-dwelling Older Adults With Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geriatric Education and Research Institute (Other Government)
Responsible Party: Principal Investigator, Tou Nien Xiang, Research Fellow, Geriatric Education and Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GERI1640
Record Dates: First submitted 2025-08-05; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Dementia
Keywords: Dementia; Resistance training; Exercise
MeSH Terms: conditions — Dementia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Quasi-experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive resistance training (Experimental): Participants in the intervention arm will receive a 16-week progressive resistance training programme implemented by center staff in a community dementia daycare center.
  Interventions: Other: Minimal-equipment progressive resistance training
- Usual Care (No Intervention): Participants in the control arm will continue receiving the usual care provided at the community dementia daycare center.

INTERVENTIONS:
Other: Minimal-equipment progressive resistance training — The intervention consists of resistance training exercises that target major upper and lower body muscle groups with the use of portable equipment such as resistance bands and wrist/ankle weights. The exercise dosage will be progressively increased across the 16 weeks to achieve training adaptations. The exercise programme will be conducted three times per week, with each session lasting approximately 30 to 45 minutes.
  Arms: Progressive resistance training

SUMMARY:
The aim for this study is to investigate the effectiveness of a 16-week minimal-equipment progressive resistance training program compared to usual care, in improving functional outcomes among older adults with dementia in Singapore.

Participants will:

* receive either minimal-equipment progressive resistance training or continue with usual care
* perform physical and cognitive function tests at three time-points

ELIGIBILITY:
Inclusion Criteria:

* Aged 55 years or older
* Community-dwelling
* Formal medical diagnosis of dementia of any cause

Exclusion Criteria:

* Diagnosis of neurological and/or myopathic disorders
* Severe audio-visual impairment
* Severe mobility impairment that affects study participation
* Not suitable to participate in exercise intervention as deemed by a nursing staff or allied health professional

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in handgrip strength | Baseline, Mid-intervention (Week 9), Post-intervention (Week 17)
  This test is a measurement of upper limb strength. Handgrip strength will be measured in kilograms using a Jamar Plus + Digital Hand Dynamometer. Participants will squeeze the dynamometer with maximum effort in a seated position with their arms at their sides and elbows flexed at 90 degrees. Two trials will be administered for each arm and the highest of four readings will be used for analysis.
Change in five times sit-to-stand test | Baseline, Mid-intervention (Week 9), Post-intervention (Week 17)
  This test is a measurement of lower limb strength. Participants will be instructed to perform five chair stands as fast as possible using a chair without arms, and the time recorded will be used for analysis.
Change in 30-seconds sit-to-stand test | Baseline, Mid-intervention (Week 9), Post-intervention (Week 17)
  This test is a measurement of lower limb strength and power. Participants will be instructed to perform repeated chair stands as fast as possible using a chair without arms, and number of completed full stands will be recorded for analysis.

SECONDARY OUTCOMES:
Change in Time Up and Go test | Baseline, Post-intervention (Week 17)
  This test is a measurement of functional mobility. The test measures the time taken for participants to rise from a seated position, walk three metres at a comfortable speed, make a turn, walk back, and return to a seated position. Two trials will be administered, and the mean reading will be used for analysis.
Change in Short Physical Performance Battery test | Baseline, Post-intervention (Week 17)
  This test is a measurement of physical function that consists of three components inclusive of 4-metre gait speed test, five times sit-to-stand test and a progressive test of standing balance.
Change in gait speed test | Baseline, Post-intervention (Week 17)
  The test measures the time taken for participants to walk six metres at a normal pace from a moving start without deceleration. Two trials will be administered, and the mean reading will be used for analysis.
Change in functional reach test | Baseline, Post-intervention (Week 17)
  This test is a measurement of dynamic balance. While standing with their back to the wall, participants are instructed to reach forward with their dominant arm outstretched at shoulder level while maintaining a fixed stance. The distance between the metacarpal bone of the third finger in the initial position and the maximum point reached is measured. Two trials will be administered, and the better reading will be used for analysis.
Change in calf circumference | Baseline, Post-intervention (Week 17)
  This test is a surrogate measurement of muscle mass. The calf circumference is determined by the maximum value of both calves measured using a nonelastic tape.
Change in mid-upper-arm circumference | Baseline, Post-intervention (Week 17)
  This test is a surrogate measurement of muscle mass. The mid-upper-arm circumference is measured at the mid-point between the acromial surface of the scapula and the olecranon process of the elbow over the dominant arm when bent at 90 degrees using a nonelastic tape.
Change in Mini-Mental State Examination | Baseline, Post-intervention (Week 17)
  The Mini-Mental State Examination (MMSE) is a measure of global cognitive function. Participants will respond to a brief questionnaire of 11 items. The score ranges between 0 and 30. Higher scores indicate better cognitive function.
Change in Trail Making Test | Baseline, Post-intervention (Week 17)
  This is a test of cogntive function. Participants will be instructed to connect numbered and lettered circles in ascending order as quickly as possible. Time to complete the test will be recorded for analysis.
Change in EQ-5D-5L proxy index score | Baseline, Post-intervention (Week 17)
  This test is a measurement of health-related quality of life. The score ranges from -0.59 to 1 and is computed based on five dimensions with higher scores indicating better quality if life. A center staff will act as a proxy assessor on behalf of the participant.
Fall incidence | Post-intervention (Week 17)
  Number of falls sustained during intervention period.

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data will be shared along with future research publications or reports with description of all data variables.